CLINICAL TRIAL: NCT05829174
Title: Comparison of Online Group Therapy Interventions for Procrastination: A Randomized Controlled Trial With Different Cognitive Behavior Therapy (CBT) Protocols
Brief Title: Comparison of Online Group Therapy Interventions for Procrastination
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nencki Institute of Experimental Biology of the Polish Academy of Sciences (Other Government)
Collaborators: University of Social Sciences and Humanities, Warsaw (Other); Institute of Psychology, Polish Academy of Sciences (Unknown); National Science Centre, Poland (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NenckiInstitute
Record Dates: First submitted 2023-04-12; First posted 2023-04-25 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Procrastination

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Cognitive Behavioral Therapy with Techniques of Starting on Time and Planning Realistically (Experimental): 5 session (one session a week) online group therapy including several psychoeducation and cognitive modules (what is procrastination, role of rewards, work environment, belief identification, cognitive restructuring, relapse prevention) and a behavioral module: realistic planning, timely beginning.
  Interventions: Behavioral: Psychoeducation and cognitive modules; Behavioral: Behavioral module: Starting on Time and Planning Realistically
- Cognitive Behavioral Therapy with Technique of Working Time Restriction (Experimental): 5 session (one session a week) online group therapy including several psychoeducation and cognitive modules (what is procrastination, role of rewards, work environment, belief identification, cognitive restructuring, relapse prevention) and a behavioral module: working time restriction.
  Interventions: Behavioral: Psychoeducation and cognitive modules; Behavioral: Behavioral module: Working Time Restriction
- Cognitive Behavioral Intervention with Time Management Technique (Active Comparator): 5 session (one session a week) online group therapy including several psychoeducation and cognitive modules (what is procrastination, role of rewards, work environment, belief identification, cognitive restructuring, relapse prevention) and a behavioral module: pomodoro technique.
  Interventions: Behavioral: Psychoeducation and cognitive modules; Behavioral: Behavioral module: Pomodoro Time Management Technique
- Wait-list control group (No Intervention): No intervention

INTERVENTIONS:
Behavioral: Psychoeducation and cognitive modules — Psychoeducation and cognitive modules: what is procrastination, role of rewards, work environment, belief identification, cognitive restructuring, relapse prevention.
  Arms: Cognitive Behavioral Intervention with Time Management Technique; Cognitive Behavioral Therapy with Technique of Working Time Restriction; Cognitive Behavioral Therapy with Techniques of Starting on Time and Planning Realistically
Behavioral: Behavioral module: Starting on Time and Planning Realistically — Learning of realistic planning, and timely starting of work.
  Arms: Cognitive Behavioral Therapy with Techniques of Starting on Time and Planning Realistically
Behavioral: Behavioral module: Working Time Restriction — Restriction of allowed time for work, and gradual increase of allowed time, if previous time windows where effectively used.
  Arms: Cognitive Behavioral Therapy with Technique of Working Time Restriction
Behavioral: Behavioral module: Pomodoro Time Management Technique — Working in 25 minutes time intervals
  Arms: Cognitive Behavioral Intervention with Time Management Technique

SUMMARY:
The aim of this study is to compare the efficacy of two cognitive behavior therapy (CBT) protocols for procrastination with an active control protocol including cognitive-behavioral elements and with a wait-list control group. The interventions will be delivered online in group settings. All three protocols include identical psychoeducation and cognitive modules related to procrastination, but will differ in the behavioral modules. The behavioral module in one protocol is focused on starting on time and realistic planning. The second protocol implements working time restriction. The active comparator protocol implements the pomodoro time management technique. The wait-list control group will receive one of the CBT protocols after the period of waiting. It is assumed that all active conditions will be superior to the wait-list control, and that CBT protocols will be superior to the protocol including the time management technique. Primary (procrastination) and secondary (depression and anxiety) measures will be collected prior and after the interventions (or waiting period in wait-list group) and after 6-months in the three active condition groups.

ELIGIBILITY:
Inclusion Criteria:

* Bachelor's and Master's university students
* Self-reported primary difficulties related to chronic and severe procrastination
* Serious procrastination problem lasting for at least one year as confirmed during clinical interview
* Having a postponed/procrastinated project to complete in the course of therapy
* Willing to participate in the study
* Fluent in Polish language
* Computer access and stable Internet connection

Exclusion Criteria:

* Current participation in other psychotherapy
* Change of psychiatric medication during last 12 weeks
* Severe anxiety or affective disorders and any other severe psychiatric disorders that require other type of specialized care and are primary to procrastination problem (e.g. major depressive episode, social phobia, PTSD, etc.)
* Active suicidality
* Psychosis, bipolar disorder
* Alcohol or substance dependence
* Severe personality disorders (with exclusion of avoidant, dependent and obsessive-compulsive personality disorders)

Ages: 18 Years to 26 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 222 (Actual)
Dates: Start 2023-04-14 (Actual); Primary Completion 2024-06-15 (Actual); Study Completion 2024-06-15 (Actual)

PRIMARY OUTCOMES:
Change in Polish version of the Pure Procrastination Scale (PPS) | baseline assessment (week 0); mid-treatment assessment (week 3); post-treatment assessment (week 6); follow-up assessment (6 months after post-treatment assessment)
  Assessment of procrastination level. The Polish version of PPS consists of 12 items that evaluate procrastination conceptualized as a dysfunctional delay (e.g. "I am continually saying I'll do it tomorrow"; "I delay making decisions until it's too late"). Participants respond on a 5-point scale (1 = "very seldom or not true of me"; 2 = "seldom true of me"; 3 = "sometimes true of me"; 4 = "often true of me"; 5 = "very often true of true of me")
Change in Polish version of the Aitken Procrastination Inventory (API) | baseline assessment (week 0); mid-treatment assessment (week 3); post-treatment assessment (week 6); follow-up assessment (6 months after post-treatment assessment)
  Assessment of academic procrastination level. The Polish version of API consists of 19 items that evaluate the tendency of students to procrastinate in their academic tasks (e.g. "If I had an important project to do, I'd get started on it as quickly as possible", "Getting down to work often takes me a long time."). Participants respond on a 5-point scale (1 = "false"; 2 = "mostly false"; 3 = " sometimes false/sometimes true"; 4 = "mostly true"; 5 = "true").

SECONDARY OUTCOMES:
Change in Polish version of the Patient Health Questionnaire (PHQ-9) | baseline assessment (week 0); mid-treatment assessment (week 3); post-treatment assessment (week 6); follow-up assessment (6 months after post-treatment assessment)
  Assessment of depressive symptoms. The Polish version of PHQ-9 consists of 9 items that evaluate the occurrence of depressive symptoms in the last 2 weeks (e.g. "Little interest or enjoyment of your activities"). Participants respond on a 4-point Likert scale (0 = "not at all"; 1 = "on a few days"; 2 = "on more than half of the days"; 3 = "nearly every day").
Change in Polish version of the Generalized Anxiety Disorder Questionnaire-7 (GAD-7) | baseline assessment (week 0); mid-treatment assessment (week 3); post-treatment assessment (week 6); follow-up assessment (6 months after post-treatment assessment)
  Assessment of depressive symptoms. The Polish version of GAD-7 consists of 7 items that evaluate the occurrence of anxiety and excessive worry symptoms in the last 2 weeks (e.g. "Feeling afraid as if something awful might happen"). Participants respond on a 4-point Likert scale (0 = "not at all"; 1 = "on a few days"; 2 = "on more than half of the days"; 3 = "nearly every day").
Degree of completion of a particular project that the participant decided to work on during the training (e.g. a thesis, an essay, a report). | baseline assessment (week 0); mid-treatment assessment (week 3); post-treatment assessment (week 6)
  Before and after therapy participants will be asked to assess the degree of completion of this project in percents.

OTHER OUTCOMES:
Change in Polish version of the subscales Low work discipline and Fear of failure of the Study Problems Questionnaire (SPQ) | baseline assessment (week 0) mid-treatment assessment (week 3);; post-treatment assessment (week 6); follow-up assessment (6 months after post-treatment assessment)
Change in Polish version of the Sensitivity to Punishment and Sensitivity to Reward Questionnaire - Short Form (SPSRQ-SF) | baseline assessment (week 0); mid-treatment assessment (week 3); post-treatment assessment (week 6); follow-up assessment (6 months after post-treatment assessment)
Change in Polish version of the Multidimensional-Multiattributional Causality Scale (MMCS) | baseline assessment (week 0); mid-treatment assessment (week 3); post-treatment assessment (week 6); follow-up assessment (6 months after post-treatment assessment)
Change in Polish version of the Performance Failure Appraisal Inventory (PFAI) | baseline assessment (week 0); mid-treatment assessment (week 3); post-treatment assessment (week 6); follow-up assessment (6 months after post-treatment assessment)
Change in Polish version of the Difficulties in Emotion Regulation questionnaire (DERS) | baseline assessment (week 0); mid-treatment assessment (week 3); post-treatment assessment (week 6); follow-up assessment (6 months after post-treatment assessment)
Change in Polish version of the Motivation Diagnostic Test (MDT) | baseline assessment (week 0); mid-treatment assessment (week 3); post-treatment assessment (week 6); follow-up assessment (6 months after post-treatment assessment)
Change in Polish version of the Zimbardo Time Perspective Inventory | baseline assessment (week 0); mid-treatment assessment (week 3); post-treatment assessment (week 6); follow-up assessment (6 months after post-treatment assessment)
Change in Polish version of the Metacognitive Beliefs about Procrastination Questionnaire (MBPQ) | baseline assessment (week 0); mid-treatment assessment (week 3); post-treatment assessment (week 6); follow-up assessment (6 months after post-treatment assessment)
Change in Polish version of the Impulsivity Scale (UPPS-P) | baseline assessment (week 0); mid-treatment assessment (week 3); post-treatment assessment (week 6); follow-up assessment (6 months after post-treatment assessment)
Change in Polish version of the Self-control Scale (NAS-50) | baseline assessment (week 0), mid-treatment assessment (week 3), post-treatment assessment (week 6), follow-up assessment (6 months after post-treatment assessment)
Change in Polish version of Positive and Negative Affect Schedule (PANAS) in relation to a project that the participant decided to work on during the training (e.g. a thesis, an essay, a report) | baseline assessment (week 0), mid-treatment assessment (week 3), post-treatment assessment (week 6)
Polish version of the Group Session Rating Scale (GSRS) | During the treatment (after each therapy session - weeks 1-5)
Polish version of the Credibility Expectancy Questionnaire (CEQ) | After the first session (week 1)
Polish version of the Negative Effects Questionnaire (NEQ) | Post-treatment (week 6)
Polish version of the Client Satisfaction Questionnaire (CSQ) | Post-treatment (week 6)

CONTACTS AND LOCATIONS:
Overall Officials: Marek Wypych, PhD, DSc, Principal Investigator — Nencki Institute of Experimental Biology, Polish Academy of Sciences; Jarosław Michałowski, Prof., Principal Investigator — SWPS University of Social Sciences and Humanities; Joachim Kowalski, PhD, Principal Investigator — Institute of Psychology, Polish Academy of Sciences
Locations (1):
- Nencki Institute of Experimental Biology, Polish Academy of Sciences, Warsaw, Poland